CLINICAL TRIAL: NCT04740671
Title: A Phase 3, Randomized, Double-masked, Active Controlled Study to Compare the Efficacy and Safety of HLX04-O Administered by Intravitreal Injection with Ranibizumab in Subjects with Wet Age-related Macular Degeneration (wAMD)
Brief Title: A Phase 3 Study to Compare the Efficacy and Safety of HLX04-O with Ranibizumab in Subjects with WAMD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HLX04-O-wAMD
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Age Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- HLX04-O (Experimental): Biologic recombinant anti-VEGF humanized monoclonal antibody
  Interventions: Drug: HLX04-O
- Ranibizumab (Active Comparator): Biologic anti-VEGF recombinant humanized monoclonal antibody fragment
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: HLX04-O — Biologic recombinant anti-VEGF humanized monoclonal antibody, developed by Shanghai Henlius Biotech, Inc.
  Arms: HLX04-O
Drug: ranibizumab — Biologic anti-VEGF recombinant humanized monoclonal antibody fragment
  Arms: Ranibizumab

SUMMARY:
This study will compare the efficacy and safety of HLX04-O administered by intravitreal injection (IVT) with ranibizumab in patients with active wAMD.

DETAILED DESCRIPTION:
This is a Phase 3, Randomized, Double-masked, Active Controlled Study to Compare the Efficacy and Safety of HLX04-O Administered by Intravitreal Injection with Ranibizumab in Subjects with wet Age-related Macular Degeneration (wAMD). This study will be conducted in approximately 90 sites in different countries or regions.

ELIGIBILITY:
Inclusion Criteria:

1. Capable to understand and sign the informed consent form (ICF) which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.
2. Women or men aged ≥50 years when signing the ICF.
3. In the Investigator's judgment, willing and able to complete all visits and assessments adhering to the prohibitions and restrictions specified in this protocol.
4. Newly diagnosed, untreated, active CNV lesions secondary to age-related macular degeneration that affect the central subfield (CSF) in the study eye. Active CNV was defined as leakage on fluorescein angiography (FA) and subretinal or intraretinal fluid on optical coherence tomography (OCT) with confirmation of the reading center during screening.
5. The total lesion area (including hemorrhage, scar and neovascularization) of the study eye ≤12 disc area (DA) with confirmation of the reading center before randomization
6. The BCVA letters between 24 and 73, inclusive, in the study eye, using Early Treatment Diabetic Retinopathy Study (ETDRS) charts.
7. Participants' fellow (non-study) eye must have a BCVA of 24 letters or better.
8. Clear ocular media and adequate pupillary dilatation to allow acquisition of good quality retinal images to confirm the diagnosis.

Exclusion Criteria:

1. Macular-related retinal pigment epithelial tears in the study eye; scar, fibrosis or atrophy involving the fovea, or CNV due to other causes in the study eye (e.g., ocular histoplasmosis, trauma,pathological myopia, etc.) with confirmation of the reading center.
2. The fellow (non-study) eye needs anti-VEGF IVT injection (e.g. CNV due to wAMD, trauma, pathological myopia, retina vein occlusion, diabetic macular edema, etc.) in the next 3 months after randomization, in the investigator's judgment.
3. Aphakia (except intraocular lens) or posterior capsular rupture of the lens (except yttrium-aluminium-garnet (YAG) laser posterior capsulotomy after intraocular lens implantation ≥30 days prior to first dose) in the study eye.
4. Active or recent (within 1 month prior to dose 1) intraocular, extraocular or periocular infection (including conjunctivitis, keratitis, scleritis or endophthalmitis), or history of idiopathic or autoimmune-associated uveitis in either eye.
5. Vitreous hemorrhage in the study eye within 3 months prior to dose 1.
6. Corneal dystrophy or history of corneal transplantation, scleral softening or history of scleral softening, history of rhegmatogenous retinal detachment or macular hole (Stage II, III or IV) in the study eye.
7. Uncontrolled glaucoma in the study eye (defined as intraocular pressure [IOP] ≥25 mmHg despite treatment with antiglaucoma medication), and/or glaucoma filtering surgery (e.g., trabeculectomy, scleral nipping, non-penetrating trabeculectomy, etc.)
8. Equivalent spherical diopter of the study eye ≥-8D. For participants who had undergone refractive correction or cataract surgery, the equivalent spherical diopter of the study eye before surgery ≥-8D.
9. Estimated by the Investigator, any concurrent intraocular condition except wAMD (e.g., diabetic retinopathy, dry AMD, retina vein occlusion, uveitis, angioid streaks, retinal detachment, epiretinal membrane, amblyopia, central serous chorioretinopathy, etc.) in the study eye that limited the potential to gain visual acuity upon treatment with the investigational product, or could have required medical or surgical intervention during the study to prevent or treat visual loss.
10. Underwent intraocular surgery including verteporfin photodynamic therapy (PDT), transpupillary thermotherapy, macular translocation, vitrectomy, laser photocoagulation in macular area, other surgery in macular area or surgery to treat AMD.
11. Previous extraocular or periocular surgery within 1 month or intraocular surgery (except the surgery mentioned in exclusion 10 ,such as cataract surgery, etc.) within 3 months prior to dose 1, or current unhealed wound, moderate or severe ulcer or fracture in the study eye.
12. Subconjunctival or intraocular use of corticosteroids within 3 months (including subconjunctival or intraocular long-acting implant within 6 months) prior to dose 1 in the study eye. Use of systemic corticosteroids for 30 or more consecutive days within 3 months prior to dose 1. Inhaled, nasal or dermal steroids are permitted. Topical ocular corticosteroids administered for 30 or more consecutive days in the study eye within 3 months prior to dose 1.
13. Previous systemic anti-VEGF therapy or IVT injection of any anti-VEGF drug into either eye or other ocular use of anti-VEGF drug within 3 months prior to dose 1.
14. Participated in any drug (other than vitamins and minerals) or device clinical trials 3 months or the duration of 5 half-lives of the study drug (which is longer) before the first dose and have used the test drug or received device treatment.
15. Pregnancy or lactation, or fertile men or women not willing to use effective contraception from the day when ICF was signed to at least 6 months following the last dose of study intervention.
16. Infertile women or men fail to meet either of the following ones: 1) menopause (≥12 continuous months of amenorrhea with no identified cause other than menopause before screening); 2) surgically sterilized.

    Fertile women or men fail to meet either of the following ones: 1) women of childbearing potential must have a negative urine or serum pregnancy test result within 14 days prior to initiation of the study intervention, and should not breastfeed. If the urine pregnancy test is positive, it must be confirmed by a serum pregnancy test; 2) agreement to remain abstinent (refrain from heterosexual intercourse) or use effective contraceptive methods from signed ICF to at least 6 months following the last dose of study intervention. Effective contraceptive methods with a failure rate of <1% per year, including bilateral tubal ligation, male sterilization, established, proper use of hormonal contraceptives that inhibit ovulation, hormone releasing intrauterine devices (IUDs), and copper IUDs.
17. In the Investigator's judgment, there is evidence of a disease or condition that contraindicates the use an investigational drug or that might affect interpretation of the results of the study or render the participant at high risk for treatment complications (e.g. stroke or myocardial infarction within 6 months prior to dose 1, uncontrolled hypertension (systolic blood pressure ≥160 mmHg, or diastolic blood pressure ≥100 mmHg), etc.).
18. Uncontrolled diabetes (defined as HbA1c>10.0%).
19. Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) is more than twice the upper limit of normal (ULN), and/or serum creatinine is 1.2 times more than the ULN, and is clinically significant in the opinion of the Investigator.
20. Abnormal coagulation function: prothrombin time(PT) or International normalized ratio (INR) ≥ 1.5 ×ULN, or activated partial thromboplastin time (aPTT) ≥1.5 ×ULN, and is clinically significant in the opinion of the Investigator.
21. Active disseminated intravascular coagulation and obvious bleeding tendency within 3 months prior to dose 1.
22. Evidence of significant uncontrolled concomitant diseases such as cardiovascular diseases, nervous system diseases, respiratory system diseases, urinary system diseases, digestive system diseases and endocrine diseases (e.g., stroke, myocardial infarction).
23. Current treatment for active systemic infection, or history of recurrent serious infections.
24. Known active or suspected autoimmune diseases, requiring systemic immunosuppressive therapy.
25. Positive for syphilis screening test human immunodeficiency virus (HIV) infection or positive for HIV screening test.
26. Known allergy to any component of the study intervention or history of allergy to fluorescein or indocyanine green, any anesthetics or antimicrobial agents used during the course of the study.
27. In the Investigator's judgment, other conditions considered not amenable to this study.
28. Participant who has been diagnosed to be COVID-19 within 2weeks prior to the first dose, or still symptomatic from an earlier infection (except symptoms associated with "Long COVID "), or displaying symptoms consistent with COVID-19 in the absence of a confirmed Covid-19 infection.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in BCVA at at Week 36 | up to at Week 36
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan

SECONDARY OUTCOMES:
Key Secondary Outcome : Mean change from baseline in BCVA at Week 48. | up to Week 48
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Mean change in BCVA over time | up to Week 48
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Proportion of patients gaining at least 15 letters in the BCVA at Week 12, 24, 36 and 48 | up to Week 12, 24, 36 and 48
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Proportion of patients gaining at least 10 letters in the BCVA at Week 12, 24, 36 and 48 | up to Week 12, 24, 36 and 48
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Proportion of patients gaining at least 5 letters in the BCVA at Week 12, 24, 36 and 48 | up to Week 12, 24, 36 and 48
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
• Mean change from baseline in size of CNV and total area of fluorescein leakage from CNV on FA at Week 12, 36 and 48 (as measured by the Reading Center) | up to Week 12, 36 and 48
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
• Mean change from baseline in CRT on OCT at Week 12, 24, 36 and 48 (as measured by the Reading Center) | up to week 12, 24, 36 and 48
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan
Change from baseline in NEI VFQ-25 scale score at Week 12, 36, and 48. | up to Week 12, 36, and 48
  Detailed Outcome Measure will be defined in the Statistical Analysis Plan

CONTACTS AND LOCATIONS:
Locations (126):
- United States (42):
  - Associated Retina Consultants-Gilbert, Gilbert, Arizona
  - Associated Retina Consultants-Phoenix, Phoenix, Arizona
  - Retina Consultants of Orange County, Fullerton, California
  - Global Research Management, Glendale, California
  - Atlantis Eyecare, VMR Institute, Huntington Beach, California
  - VMR Institute, Huntington Beach, California
  - South Coast Retina Center, Long Beach, California
  - Retina Consultants of Orange County, Los Alamitos, California
  - MACRO Trials/ Lazar Retina, Los Angeles, California
  - East West Eye Institute, Torrance, California
  - Retina Consultants of Southern Colorado, Colorado Springs, Colorado
  - Florida Retina Institute-Orlando, Jacksonville, Florida
  - Florida Retina Institute-Orlando, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - Southeast Retina Center, Augusta, Georgia
  - The University of Chicago, IL, Chicago, Illinois
  - The University of Chicago, Chicago, Illinois
  - Illinois Retina Associates, Oak Park, Illinois
  - Retina Associates LLC, Lenexa, Kansas
  - Butchertown Clinical Trials, Louisville, Kentucky
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Retina Consultants of Minnesota, Edina, Minnesota
  - VitreoRetinal Surgery PLLC DBA Retina Consultants of Minnesota, Saint Louis Park, Minnesota
  - Mississippi Retina Associates, Jackson, Mississippi
  - Piedmont Retina Specialists, Asheville, North Carolina
  - Western Carolina Retinal Associates, Asheville, North Carolina
  - Graystone Eye, Hickory, North Carolina
  - North Carolina Retina Associates, Wake Forest, North Carolina
  - Verum Research, LLC, Eugene, Oregon
  - Retina Consultants of Charleston - Beaufort, Beaufort, South Carolina
  - Retina Consultants of Charleston: Charleston Neuroscience Institute, Charleston, South Carolina
  - Carolina Center for Sight, Florence, South Carolina
  - Retina Consultants of Nashville, Nashville, Tennessee
  - Retina Consultants of TEXAS- Newcastle, Bellaire, Texas
  - Mt. Olympus Research-Garcia, Houston, Texas
  - Mt. Olympus Research/Museum Eye District, Houston, Texas
  - Retina Consultants of TEXAS - Round Rock, Round Rock, Texas
  - Retina Consultants of Texas, The Woodlands, Texas
  - Retina Associates of Utah, PLLC, Salt Lake City, Utah
  - Rocky Mountain Retina Consultants, Salt Lake City, Utah
  - Emerson Clinical Research Institute, Falls Church, Virginia
- Australia (3):
  - Lions Eye Institute, Nedlands, Western Australia
  - The Alfred Hospital, Melbourne
  - Lions Eye Institute, Nedlands
- Bulgaria (10):
  - Mhat Dr. Stamen Iliev Ad, Montana, Montana
  - Assoc. Prof. Dr. Desislava Koleva Aipsmaed Sveti Luka Eood, Plovdiv, Plovdiv
  - Dcc Aleksandrovska Eood, Sofia, Sofia
  - Umhat Lozenets Ead, Sofia, Sofia
  - University First Mhat - Sofia Sv. Joan Krastitel Ead, Sofia, Sofia
  - Specialized Hospital For Active Treatment in Ophthalmology - Varna, Varna, Varna
  - Vizus Eood, Gorna Oryahovitsa, Veliko Tarnovo
  - Specialized Eye Hospital For Active Treatment - Burgas Ltd, Burgas
  - Medical Center Dar Plovdiv Ltd, Plovdiv
  - Medical Center Vereya Ltd, Stara Zagora
- China (8):
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Joint Shangtou International Eye Center Of Shantou University And The Chinese University Of Hong Kong, Shantou, Guangdong
  - The Third Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - First Hospital of Jilin University, Changchun, Jilin
  - The People's Hospital of Ningxia Hui Autonomous Region, Yinchuan, Ningxia
  - Weifang Eye Hospital, Weifang, Shandong
  - Shanghai First Peoples's Hospital, Shanghai, Shanghai Municipality
  - Shanxi Eye Hospital, Taiyuan, Shanxi
- Oftex Ocni Klinika, Pardubice, Czechia
- France (2):
  - Centre Hospitalier Universitaire Amiens-Picardie Service D'Ophthalmologie Amiens France, Amiens
  - University Eye Clinic Centre Hospitalier Creteil Paris France, Paris
- Germany (6):
  - Ukb University of Bonn, Bonn
  - University Hospital Freiburg, Freiburg im Breisgau
  - Justus Liebig University Giessen, Giessen
  - Johannes Gutenberg University Mainz, Mainz
  - St Franziskus Hospital Munster, Münster
  - Eye Clinic Sulzbach, Sulzbach
- Hungary (6):
  - Bajcsy-Zsilinszky Korhaz Es Rendelointezet, Budapest, Budapest
  - Semmelweis Egyetem, Budapest
  - Markhot Ferenc Oktatokorhaz Es Rendelointezet, Eger
  - Ganglion Orvosi Kozpont, Pécs
  - Pecsi Tudomanyegyetem Klinikai Kozpont - Szemeszeti Klinika, Pécs
  - Szegedi Tudomanyegyetem Aok Szakk, Szeged
- Italy (4):
  - Irccs Fondazione G.B. Bietti Per Lo Studio E La Ricerca in Oftalmologia Onlus Rome, Italy, Rome, Rome
  - Clinica Oculistica Ospedale Luigi Sacco, Universita' Degli Studi Di Milano, Milan
  - Clinica Oculistica Universita Vita Salute - Irccs Ospedale San Raffaele, Milan
  - Fondazione Policlinico Universitario Agostino Gemelli - Irccs Uoc Oculistica, Rome
- Latvia (2):
  - P Stradina Clinical University Hospital, Riga
  - Riga East University Hospital, Riga
- Poland (12):
  - Nzoz E-Vita, Bialystok, Podlaskie Voivodeship
  - Centrum Medyczne Promed, Krakow, WA
  - Oftalmika Sp Z.O.O, Bydgoszcz
  - Centrum Klinicke Oftalmologie S.R.O, Katowice
  - Szpital SW. Rozy, Krakow
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 W Lubline, Lublin
  - Szpital SW Wojciecha, Poznan
  - Caminomed Wojciech Jedrzejewski, Tarnowskie Góry
  - Centrum Medyczne Uno-Med, Tarnów
  - Nzoz Optimed, Warsaw
  - Retina Okulistyka Sp.Z O.O.Sp.K., Warsaw
  - Centrum Medyczne Piasta 47, Wałbrzych
- Serbia (2):
  - Special Optalmological Hospital Belgrade, Belgrade
  - Zvezdara University Medical Center, Belgrade
- National University Hospital, Singapore, Singapore
- Slovakia (7):
  - Ocna Klinika Szu F.D.R.Banska Bystrica, Banská Bystrica
  - Fakultna Nemocnica Nitra, Nitra
  - Fakultna Nemocnica S Poliklinikou Nove Zamky Oftalmologicke Nelozkove Oddelenie, Nové Zámky
  - Nemocnica Poprad As Oftalmologicke Oddelenie Jzs, Poprad
  - Nemocnica S Poliklinikou Trebisov A.S. Ocne Oddelenie Jzs, Trebišov
  - Fakultna Nemocnica Trencin, Trenčianske Teplice
  - Fakultna Nemocnica S Poliklinikou Zilina, Žilina
- Spain (20):
  - VISSUM, Alicante
  - Centro de Oftalmologia Barraquer, Barcelona
  - Hospital Universitari Vall D Hebron, Barcelona
  - Institito de Microcirugia Ocular, Barcelona
  - Institut Catala de La Retina, Barcelona
  - Oftalvist Clinic, Burjassot
  - Hospital La Arruzafa, Córdoba
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda
  - Instituto Oftalmologico Fernandez-Vega, Oviedo
  - Clinica Universitario de Navarra, Pamplona
  - Hospital Universitario Donostia, San Sebastián
  - Omiq Hospital General de Catalunya, Sant Cugat del Vallès
  - Hospital Universitario Virgen Macarena, Seville
  - Clinica Oftalmologica Aiken, Valencia
  - Consorcio Hospital General Universitario de Valencia, Valencia
  - Fisabio Oftalmologia Medica, Valencia
  - Hospital Rio Hortega, Valladolid
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No